## Informed Consent Addendum

NCT04175106

Date: 04-Aug-2020



Participant Printed Name



## Informed Consent Addendum Research During COVID-19 Pandemic

These research activities are taking place during the COVID-19 Pandemic. The researchers involved in this study have no symptoms of COVID-19 and have not knowingly interacted with anyone demonstrating symptoms or diagnosed as COVID-19 positive.

The sanitation and cleaning measures in place during all study activities are: sanitation of participant and staff accessed areas with 70% alcohol solution before and between use by researchers and each participant, with limited access to procedure areas by participants and outside staff, and hand washing with soap and water before direct contact with researchers, participants, equipment and high touch surfaces. The personal protective equipment (PPE) that the researchers will use includes masks, face shields, gowns and gloves. Gloves will be changed after each participant. As a participant, you will be provided a mask as PPE and you must wear it while participating in this research.

## Participants, Please Initial I have not knowingly interacted with someone who has been diagnosed or demonstrated symptoms of COVID-19 I do not have any symptoms of COVID-19 such as cough, fever, shortness of breath, chills, muscle pain, new loss of taste or smell. I agree to follow all safety and sanitation procedures while participating in this study including wearing appropriate personal protective equipment. I understand that though all of these safety measures are put in place to protect my health as a participant, there is a risk that I may still transmit or contract COVID-19. There is no provision for compensation or free medical care for me if I contract or transmit COVID-19 as a result of my participation in this study. • I understand that in order to take part in this research, while I am a participant in this study I must allow my name and information about those I interacted with to be recorded for contact tracing purposes should an issue arise regarding COVID-19 infection or transmission. I have read the above information and have had the opportunity to ask questions and have them answered. I understand my responsibility related to COVID-19 and and the risks associated with being in this study as a result. I agree to participate in this research.

Participant Signature

Date